CLINICAL TRIAL: NCT02076516
Title: Pilot Evaluation Of CORACTO® (Rapamycin-Eluting Coronary Stent Delivery System) in The Treatment Of Patients With Coronary Artery Disease
Brief Title: Pilot Evaluation Of CORACTO® (THE PILOT-SECRET TRIAL)
Acronym: PILOT-SECRET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alvimedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALV-01
Record Dates: First submitted 2014-02-28; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Disease
Keywords: Drug-eluting Stent,Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug-eluting stent: CORACTO® (Experimental): Single arrm
  Interventions: Device: Drug-eluting stent: CORACTO®

INTERVENTIONS:
Device: Drug-eluting stent: CORACTO®

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the CORACTO® (Rapamycin®-Eluting coronary stent delivery system) for the treatment of up to two de novo lesions or restenotic post-PTCA (non-stented) lesions located in up to two epicardial native coronary arteries (maximum one lesion per vessel) suitable for treatment with stents from 2.5 to 4.0 mm in diameter < than 15 mm suitable for treatment with a single CORACTO® stent in a population of 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old.
* Patient is eligible for percutaneous coronary intervention (PCI) and acceptable candidate for coronary artery bypass grafting (CABG).
* Clinical evidence of ischemic heart disease and/or a positive functional study, stable angina pectoris (Canadian Cardiovascular Society Classification (CCS) 1, 2, 3 or 4) or unstable angina pectoris (Braunwald Class IB-C, IIB-C, or IIIB-C), or silent ischemia.
* The target lesion(s) or target vessel(s) meet(s) all the following criteria:

  1. The target lesion is a single de novo lesion in a native coronary artery.
  2. The stenosis of target lesion(s) is ≥ 50% and < 100% (by visual estimation).
  3. The target lesion length must be ≤ 15 mm. In case that a second stent should be required for successful treatment, it should be a CORACTO® stent.
  4. The target reference vessel diameter must be (by visual estimation) suitable for treatment with stents between 2.5 and 4.0 mm.
* Patient has been informed of the nature of the study, understands the study requirements, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site.
* The patient is willing and able to comply with all specified follow-up evaluations.

Exclusion Criteria:

* Most recent left ventricular ejection fraction (LVEF) of the patient is < 25%.
* Known allergies to the following: aspirin, Clopidogrel bisulfate (Plavix®), Prasugrel (Effient®) or Ticlopidine (Ticlid®), heparin, Rapamycin, stainless steel, Poly Lactic - co- glycolic acid or contrast agent (that cannot be adequately premedicated).
* Platelet count is less than 100,000 cells/mm3 or more than 700,000 cells/mm3.
* White Blood Cell count is less than 3,500 cells/mm3.
* Evidence of an ST-segment elevation acute myocardial infarction (MI) or non-ST segment elevation MI with positive Troponin within 72 hours before the intended treatment.
* ANY previous PCI
* Planned staged procedures (patient with 2-vessel disease should be treated during the same procedure). Presence of any other significant lesion of > 50% stenosis (by visual estimation) anywhere within the target vessel
* Significant lesions in any non-target vessel that will require interventional treatment within 30 days post-procedure
* Planned future interventional procedure in the target vessel .
* The target lesion(s) require(s) treatment with a device other than PTCA balloon prior to stent placement. (e.g. but not limited to directional coronary atherectomy, excimer laser, rotational atherectomy, thrombus aspiration etc.).
* Previous stenting anywhere within the target vessel(s)
* Target vessel has evidence of thrombus
* Excessive tortuosity (> 60°) of the target vessel proximal to the target lesion (by visual estimation).
* The target lesion(s) has any of the following characteristics (by visual estimation):

  1. Ostial or bifurcation lesion (within 3mm from region of origin of target vessel, by visual estimation).
  2. Target lesion involves a side branch > 2mm in diameter.
  3. Moderate to severely calcified lesion which cannot be successfully predilated.
  4. Target lesion is located in or supplied by an arterial or venous bypass graft.
  5. A complete occlusion (TIMI flow 0 or 1).
* Target lesion is located in left main trunk.
* Stroke or transient ischemic attack within 180 days prior to the baseline procedure.
* Active peptic ulcer or upper GI bleeding within 180 days prior to the baseline procedure.
* The patient has bleeding haemorrhagic diathesis or coagulopathy.
* The patient will refuse a blood transfusion.
* The patient has a widespread peripheral vascular disease.
* Acute or chronic renal dysfunction (creatinine clearance below 40ml/m2).
* The patient requires multiple stent implantations for a tandem lesion.
* Life expectancy less than 1 year.
* Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
* In the Investigator's opinion patient has (a) co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.
* Female of childbearing potential, pregnant and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
In-stent late loss (LL) in patients implanted with a CORACTO® stent (per protocol analysis) | at 6 months

SECONDARY OUTCOMES:
Stent Thrombosis ( Definite and probable) | at 30 days, 6 months and 12 months

OTHER OUTCOMES:
Device-oriented Target Lesion Failure (TLF) | at 30 days, 6 months and 12 months
  Device-oriented Target Lesion Failure (TLF) defined as the composite of Cardiac Death, Target Vessel Myocardial Infarction (TV-MI), Clinically indicated Target lesion Revascularization (CI-TLR)
Patient Oriented Composite Endpoint Major Adverse Cardiac Events (MACE) | at 30 days, 6 months and 12 months
  Patient Oriented Composite Endpoint Major Adverse Cardiac Events (MACE) defined as any cause mortality, Myocardial Infarction MI (Q-wave and non-Q-wave) or any clinically indicated Target Vessel Revascularization
Total Revascularization Rate (clinically and non-clinically driven) | at 30 days, 6months and 12 months
Percentage of uncovered struts at Follow Up (as measured at FU Optical Coherence Tomography (OCT) imaging) | at 6 months
Late-appearing stent malapposition (as documented from post- and FU Optical Coherence Tomography (OCT) imaging and expressed both as dichotomous and continuous manner [number / percentage of late-appearing malapposed struts]) | at 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- ZNA Middleheim, Antwerp, Belgium
- France (2):
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Hospital Prive Jacques Cartier, Massy
- Hospital Clínico San Carlos, Madrid, Spain
- Bezmialem University Hospital, Istanbul, Turkey (Türkiye)